CLINICAL TRIAL: NCT03338140
Title: Assistant Lecturer of Urology in Assiut University
Brief Title: Outcome of Living Donor Renal Transplantation in Assiut Urology and Nephrology University Hospital ,Initial Experience
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Mostafa Abdel Gawad, Assistant lecturer, Assiut University
Other Study IDs: Renal transplantation
Record Dates: First submitted 2017-10-23; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Renal Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
evaluation of outcome of living donor renal transplantation in assiut urology and nephrology university Hospital regarding the survival of patients and grafts , complications and quality of life after transplantation.

DETAILED DESCRIPTION:
Renal failure is a widespread life threatening problem affecting a variety of age groups that needs a replacement therapy either regular dialysis with its drawbacks or kidney transplantation. Kidney transplantation is the treatment of choice for suitable candidates with ESRD. Since the advent of kidney transplantation in 1954, allograft and patient survival in the world have markedly improved because of advances in surgical techniques and immunosuppression. Few studies have compared kidney transplant outcomes In different countries. Because of varying allocation policies, cultural differences influencing preferences for living vs deceased donation, and government-funded health care in some countries, it is possible that post transplant outcomes are vastly different in other countries. Many studies described the current status of kidney allograft and patient survival in different countries based on data from the 2014 Scientific Registry of Transplant Recipients (SRTR) Annual Data Report. These outcomes are compared with those from Australia and New Zealand (ANZ), Europe, and Canada, using the most recent published registry data. A study was conducted showing that a total of 17,814 adult kidney transplants were performed in the United States in 2014. Of these, 12,279 were from deceased donors and 5535 were from living donors. Deceased donor allograft survival rates have improved over time. The most recent SRTR annual report showed long-term outcome data on recipients who underwent transplant from 1991 to 2014. From 2010 to 2014, the unadjusted 1-year allograft survival rate for recipients of a first deceased donor kidney transplant was 93.4% . For second or subsequent deceased donor transplants, the 1- year unadjusted allograft survival rate was comparable at 92.5%. It is well established that living donor kidney transplants are associated with superior post-transplant outcomes compared with deceased donor transplants, and this was reflected in the SRTR data. In recipients undergoing a primary living donor kidney transplant, the 1-year unadjusted allograft survival rate was 97.2%. In those undergoing retransplant from a living donor (first transplant from deceased or living donor), 1-year allograft survival was similar at 97.3%. Five-year unadjusted allograft survival rates for a first living donor kidney transplant and a second or subsequent transplant were 84.6% and 81.4%, respectively. Despite better outcomes, numbers of living donor transplants in the United States have decreased over the past 10 years; the largest decrease was in living-related donor kidney transplants, from 4340 in 2004 to 2693 in 2014.This underscores the ongoing need to encourage and support living donation. Potential explanations for the decline in living kidney donation include an aging U.S.A population such that potential donors are older, often have more comorbidity, and may not be medically suitable, financial disincentives, changes in organ allocation and donor selection criteria, and inadequate public awareness about the benefits of living organ donation.Although the recipient's health insurance covers the donor's donation related medical expenses, it does not reimburse for other expenses (eg, travel to the transplant center for predonation testing and surgery, lodging, lost wages during the post-surgery recovery period, especially for selfemployed or part-time workers, and higher premiums for health or life insurance or, difficulty obtaining it, after donation).The average out-of-pocket cost incurred by patients after living donation is reported to be $5000. In June 2014, the transplant community convened a Consensus Conference on Best Practices in Live Kidney Donation and issued several recommendations with the goal of making living donation financially neutral. Progress is being made as the Living Donor Protection Act was introduced in Congress in February 2016. A study showed that Patient Survival Recipients of living donor kidney transplants enjoy high survival rates, with little difference in outcomes for primary transplant and retransplant. The unadjusted 1-year patient survival rate was 97.0% for primary deceased donor transplant recipients from 2010 to 2014 and 97.2% for retransplant recipients. Patient survival at 5 years was 86.1% for first-transplant recipients and 88.9% for retransplant recipients who underwent deceased donor transplant from 2005 to 2009. For living donor transplant recipients, patient survival at 1 year and 5 years was 98.7% and 93.1% (primary transplant) and 99.0% and 92.9% (retransplant), respectively. This likely reflects selection bias during the evaluation for retransplant, when patients who were non adherent (perhaps leading to allograft failure) or who have substantial comorbidity are usually not deemed candidates for retransplant. Kidney transplant before dialysis initiation is associated with better post-transplant outcomes than transplant after dialysis initiation. another study reported that less than 6 months of pretransplant dialysis was associated with a 17% higher risk of death-censored allograft loss compared with preemptive transplant. The risk of allograft loss increased with longer pre -transplant dialysis time, although the relative increase after 3 years of dialysis was minimal. Similarly, this study showed that 6 months or longer of dialysis pretransplant was linked to a higher risk of death post-transplant compared with preemptive transplant. Other advantages of preemptive transplant include lower rates of delayed graft function and lower overall ESRD treatment costs compared with maintenance dialysis. In 2014, 17.1% of U.S.A adult transplant recipients underwent a pre emptive transplant. Although the proportion of preemptive living donor transplants increased from 23% in 1995 to 32% in 2014, growth has been stagnant since 2004 despite recognition of the benefits and new paradigms, such as the Kidney First Initiative. Previously, deceased donor kidneys were classified as standard criteria donor (SCD) or expanded criteria donor (ECD). A study showed that U.S.A has the highest 1-year survival rate for both primary and retransplant cases as compared to Australia ,Canada and Europe .while Australia has the highest 5-year survival rates .Canada and Europe have the lowest survival rates.

this study will be conducted on all recipient of living donor kidney transplantation in Assiut university urology &nephrology hospital to detect the outcome regarding survival rates of both grafts & patients, post-transplant quality of life and incidence of post -transplant complications.

Survival may be short term meaning that the graft will be functioning only for the 1st year while long term survival for more than 1st year, at any time if the patient returns to regular dialysis this means failure of the graft. Quality of life will be evaluated regarding physical performance, appearance, anxiety , frustration, depression and burden of immunosuppressants , comparison between post-transplant and pre- transplant status.

Complications of renal transplantation may be surgical or non surgical . Surgical complications may be urinary as (urinary leakage,urinary obstruction, urinoma ),lymphatic (lymphocele,lymphatic leakage and lymphatic obstruction)and vascular as ( renal artery stenosis , renal vein thrombosis,vascular aneurysms and rejection) . Non surgical as ( rejection, side effects of Immunosuppressants as viral infections,nephrotoxicity,skin changes,malignancy,etc) .

ELIGIBILITY:
Inclusion Criteria:

* All recipients of renal transplantation in Assiut urology and nephrology university Hospital

Exclusion Criteria:

* All recipients of renal transplantation who were transplanted outside Assiut urology and nephrology university Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -All recipients of renal transplantation in Assiut urology and nephrology university Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of quality of life after renal transplantation | 2 years
  Evaluation of physical and physological performance changes pre and post transplantation using kidney disease quality of life(KDQOL) score

CONTACTS AND LOCATIONS:
Overall Officials: Nasreldin Abdelall, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Rodrigue JR, Schold JD, Mandelbrot DA. The decline in living kidney donation in the United States: random variation or cause for concern? Transplantation. 2013 Nov 15;96(9):767-73. doi: 10.1097/TP.0b013e318298fa61. PMID 23759882
- [Background] Tushla L, Rudow DL, Milton J, Rodrigue JR, Schold JD, Hays R; American Society of Transplantation. Living-Donor Kidney Transplantation: Reducing Financial Barriers to Live Kidney Donation--Recommendations from a Consensus Conference. Clin J Am Soc Nephrol. 2015 Sep 4;10(9):1696-702. doi: 10.2215/CJN.01000115. Epub 2015 May 22. PMID 26002904
- [Background] Clarke KS, Klarenbach S, Vlaicu S, Yang RC, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. The direct and indirect economic costs incurred by living kidney donors-a systematic review. Nephrol Dial Transplant. 2006 Jul;21(7):1952-60. doi: 10.1093/ndt/gfl069. Epub 2006 Mar 22. PMID 16554329
- [Background] Meier-Kriesche HU, Port FK, Ojo AO, Rudich SM, Hanson JA, Cibrik DM, Leichtman AB, Kaplan B. Effect of waiting time on renal transplant outcome. Kidney Int. 2000 Sep;58(3):1311-7. doi: 10.1046/j.1523-1755.2000.00287.x. PMID 10972695
- [Background] Kasiske BL, Snyder JJ, Matas AJ, Ellison MD, Gill JS, Kausz AT. Preemptive kidney transplantation: the advantage and the advantaged. J Am Soc Nephrol. 2002 May;13(5):1358-64. doi: 10.1097/01.asn.0000013295.11876.c9. PMID 11961024
- [Background] Friedewald JJ, Reese PP. The kidney-first initiative: what is the current status of preemptive transplantation? Adv Chronic Kidney Dis. 2012 Jul;19(4):252-6. doi: 10.1053/j.ackd.2012.05.001. PMID 22732045
- [Background] Rao PS, Ojo A. The alphabet soup of kidney transplantation: SCD, DCD, ECD--fundamentals for the practicing nephrologist. Clin J Am Soc Nephrol. 2009 Nov;4(11):1827-31. doi: 10.2215/CJN.02270409. Epub 2009 Sep 24. PMID 19808229